CLINICAL TRIAL: NCT00395408
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Comparing the Effect on Linear Growth of Montelukast With Placebo and Inhaled Beclomethasone in Pediatric Patients (Prepubertal, Tanner Stage I) With Mild Asthma
Brief Title: Linear Growth Study (0476-097)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-097; 2006_550
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment : 56 Weeks
Drug: Comparator : beclomethasone dipropionate / Duration of Treatment : 56 Weeks

SUMMARY:
The purpose of this study is to compare the effect of montelukast with placebo and beclomethasone on the average rate of linear growth over a period of 56 weeks in children with mild asthma.

ELIGIBILITY:
Inclusion Criteria :

* Boys (aged 6 to 8 years at Visit 1) at Tanner Stage I (prepuberty)
* Girls (aged 6 to 7 years at Visit 1) at Tanner Stage I (prepuberty
* With at least a 6-month history of asthma with typical symptoms (including, but not limited to cough, wheeze, and shortness of breath, with periodic episodes requiring treatment with inhaled beta-agonists)

Exclusion Criteria :

* Patients who used more than 2 courses of inhaled corticosteroids within the 12 months prior to Visit 1

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2000-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To establish the difference in the average rate of linear growth over the 56-week double-blind treatment period between the montelukast and placebo groups

SECONDARY OUTCOMES:
To evaluate the effects of montelukast in comparison with placebo and beclomethasone on FEV1
Beta-agonist use
Oral corticosteroid rescues for asthma
Discontinuations due to asthma
Peripheral blood eosinophil count
Markers of bone turn-over

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Becker AB, Kuznetsova O, Vermeulen J, Soto-Quiros ME, Young B, Reiss TF, Dass SB, Knorr BA; Pediatric Montelukast Linear Growth Study Group. Linear growth in prepubertal asthmatic children treated with montelukast, beclomethasone, or placebo: a 56-week randomized double-blind study. Ann Allergy Asthma Immunol. 2006 Jun;96(6):800-7. doi: 10.1016/s1081-1206(10)61342-7. PMID 16802767